CLINICAL TRIAL: NCT00773565
Title: Identification of Novel Targets for Regulation of Adipose Tissue Mass
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Gottfried Rudofsky (Other)
Collaborators: Swiss Federal Institute of Technology (Other)
Responsible Party: Sponsor-Investigator, Gottfried Rudofsky, Oberarzt, Heidelberg University
Organization: Heidelberg University (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: EFSD-CRP-2008
Record Dates: First submitted 2008-10-15; First posted 2008-10-16 (Estimated); Last update posted 2012-08-23 (Estimated); Status verified 2012-08

CONDITIONS: Obesity
Keywords: patients with obesity (BMI > 30 kg/m2)
MeSH Terms: conditions — Obesity

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Optifast (Other): Patients included take part at a weight reduction program over one year.
  Interventions: Dietary Supplement: Optifast

INTERVENTIONS:
Dietary Supplement: Optifast — Formula diet for twelve weeks combined with physical activity and behavioral therapy

SUMMARY:
The aim of this study is to understand the metabolic changes occurring in fat tissue both during controlled weight loss that lead to the improvement of type 2 diabetes and other obesity associated metabolic disorders. The novelty of the study is the analysis of preadipocytes, a poorly characterized subfraction of the adipose tissue, which provides adipocyte precursors and thereby strongly influences adipose tissue mass changes. Knowledge of pathways involved in controlling adipose tissue composition will help to design novel intervention strategies for the treatment of obesity associated metabolic disorders such as type 2 diabetes.

ELIGIBILITY:
Inclusion Criteria:

* Participants of the OPTIFAST52 program
* BMI > 30 kg/m2

Exclusion Criteria:

* Rejection of informed consent by the participant

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 62 (Actual)
Dates: Start 2008-10; Primary Completion 2011-08 (Actual); Study Completion 2011-08 (Actual)

PRIMARY OUTCOMES:
number of adipocytes and preadipocytes under weight loss | three years

SECONDARY OUTCOMES:
metabolic function of adipocytes and preadipocytes under weight loss | three years

CONTACTS AND LOCATIONS:
Overall Officials: Christian Wolfrum, PhD, Study Chair — ETH Zürich
Locations (1):
- University Hospital Heidelberg, Heidelberg, Germany